CLINICAL TRIAL: NCT06986031
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled Trial to Investigate the Efficacy and Safety of Two Concentrations of PKB171 Against Placebo in Couples With Asthenozoospermia Who With to Conceive
Brief Title: PKB171 Against Placebo in Couples With Asthenozoospermia Who Wish to Conceive
Acronym: PKB171
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was teriminated early due to low subject recruitment and high screening failure rates, despite several protocol modifications.
Sponsor: Prokrea BCN, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PKB171-02; 2016-003993-42 (EudraCT Number)
Record Dates: First submitted 2025-01-28; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-01

CONDITIONS: Infertility, Male
Keywords: Infertility, Male; asthenozoospermia; pentoxifylline
MeSH Terms: conditions — Infertility, Male; Asthenozoospermia | interventions — Menstrual Hygiene Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gel PKB171 150 mg (equivalent to 3% pentoxifylline) (Experimental): Intravaginal application of Gel PKB171 3% with a single-use applicator (syringe).
  The content of the applicator (5 g) was inserted as deep as possible into the vagina, and the female rested for at least 45 minutes in bed.
  Interventions: Drug: Vaginal product
- Gel PKB171 200 mg (equivalent to 4% pentoxifylline) (Experimental): Intravaginal application of Gel PKB171 4% with a single-use applicator (syringe).
  The content of the applicator (5 g) was inserted as deep as possible into the vagina, and the female rested for at least 45 minutes in bed.
  Interventions: Drug: Vaginal product
- Gel PKB171 placebo (Placebo Comparator): Intravaginal application of Gel PKB171 placebo with a single-use applicator (syringe).
  The content of the applicator (5 g) was inserted as deep as possible into the vagina, and the female rested for at least 45 minutes in bed.
  Interventions: Drug: Vaginal product

INTERVENTIONS:
Drug: Vaginal product — Intravaginal application of gel PKB171 with a single-use applicator (syringe)

SUMMARY:
The test medication Gel PKB171 is a vaginal gel that has not yet been licensed by the regulatory authorities. However, the active substance pentoxifylline has been available as tablets for decades and is used to increase peripheral blood flow in patients with circulation problems. Additionally, pentoxifylline is used to treat sperm samples in artificial insemination and test tube fertilisation to increase the mobility of sperm.

A first trial performed in Spain, 30 women were treated with Gel PKB171 for up to three times. Gel PKB171 was generally well tolerated and the most common side effects were local reactions like vaginal discharge and itching.

The aim of this clinical trial is to test if treatment with Gel PKB171 increases pregnancy rate in couples with reduced mobility of sperm (so-called asthenozoospermia). Additionally, the safety and local tolerability of Gel PKB171 was further investigated.

DETAILED DESCRIPTION:
Multicentre, randomised, double-blind, placebo-controlled, parallel-group trial in couples who both wish to procreate with each other. A couple consists of a male subject with asthenozoospermia and a fertile female subject.

The trial consisted of:

* a screening period (visits VS1, VS2 and VS3)
* up to three double-blind treatment cycles (Visits VR, VT1a, VTib, VT2 and VT3) and a double-blind post-treatment period (visit VP1, VP2 and VP3).

After the trial there was:

- an observation period until 32 days after delivery or termination of pregnancy (visit VP4).

Screening period:

At first visit (VS1) after giving informed consent, the couple undergo several examination to check eligibility. The trial staff interviewed the female subject to determine the usual length of ther menstrual cycle, i.. the mean value over the last six cycles.

The next visit (VS2) was performed between Day 1 and Day 5 of the female subject's mentrual cycle and after 2 to 5 days of abstinence of the male subject. The next visit (VS3) took place 12 to 15 days after VS2, and a second semen analysis will be performed.

First treatment cycle:

The next visit (VR) was performed between Day 1 and Day 5 of the female subject's next menstrual cycle. After eligibility has been confirmed, the couple was randomised to Gel PKB171 150 mg, gel PKB171 200 mg or placebo. Trial staff dispensed four units (one reserve) of IMP, ovulation test strips and subjects diary and explained their use to the couple.

Ovulation testing started 16 days before the usual end of the menstrual cycle. Therefore ovulation tests started between Day 5 and Day 19.The female was instructed to perform two ovulation tests (LH distick) each day, preferable at the same time of the day.

Within 72 hours after positive ovulation test, the couple should have three times intercourse, at intervals of 24 hours. IMP was applied after each intercourse.

Within 24 hours after second IMP, the couple attended visit VT1 for safety assessments.

The next visit (VT1B) was performed 18-20 days after positive ovulation tests of between Day 1 and Day 5 of the next menstrual cycle whatever came first.

Second treatment cycle:

If the female subject was not pregnant at VT1b trial staff dispensed IMP, ovulation test strips and subject diary for the second treatment cycle. Ovulation testing and sexual intercourse, incluidng IMP use, after positive ovulation test was repeated as in the first treatment cycle.

Visit VT2 was performed 18-20 days after positive ovulation tests of between Day 1 and Day 5 of the next menstrual cycle whatever came first.

Third treatment cycle:

If the female subject was not pregnant at VT2 trial staff dispensed IMP, ovulation test strips and subject diary for the third treatment cycle. Ovulation testing and sexual intercourse, incluidng IMP use, after positive ovulation test was repeated as in the first and second treatment cycle.

Visit VT3 was performed 18-20 days after positive ovulation tests of between Day 1 and Day 5 of the next menstrual cycle whatever came first.

Double-blind post-treatment period:

In case pregnancy was detected in the course of the trial, the next visit (VP1) was taken place 56-60 days after positive pregnancy test and fetal heart activities was examined by transvaginal ultrasound. A pregnant female subject came to visit VP2 between 8th and 16th+6 week of gestation and undergone combined first trimestre screening. The results were discussed at the next visit (VP3) which was performed up to 10 days later.

Observational period:

Within 28-32 days after delivery or termination of pregnancy. VP4 was performed, and pregnancy outcome and offspring characteristics were recorded. VP4 was performed as a telephone visit.

ELIGIBILITY:
Inclusion Criteria:

- For the couple:

1. Unable to conceive for at least 12 months, despite regular and adequate unprotected sexual intercourse.
2. Willing and able to comply with the protocol

   - For the male subjects:
3. Male subjects aged 18-50 years.
4. Two semen analyses, both with the following results:

   1. Total number of spermatozoa at least 12.000.000 per ejaculation
   2. Progressive motility less than 32%
   3. Total motility less than 40%
   4. Normal forms at least 2%
   5. Viable spermatozoa at least 45% -For the female subjects:
5. Female subjects aged 18-37 years.
6. BMI 18-30 kg/m2
7. Regular spontaneous menstrual cycles between 21 and 35 days in length (intercycle variations not more than +/- days) with the last six cycles before visit VS1.
8. Presence of both ovaries.
9. Normal uterine cavity as assessed by transvaginal sonography at VS1. No submucosal fibroids or intramural fibroids exceeding 4 cm in diameter.
10. Normal findings at hysterosalpingography. If results from within the last 24 months are available, the examination witll not be repeted at VS2.
11. AMH blood level > 1.0 ng/mL measured at VS1
12. Antral follicle count (sum of both ovaries) > 7 measured at VS2. If results the last 6 months are available, the examination will not be repeated at VS2.

Exclusion Criteria:

* For the couple:

  1. Any sexual intercourse with another partner (other than corresponding trial subject) within 12 weeks before VS1 and willing to continue until VT3.
  2. Couples who had any unsuccessful previous assisted reproductive technology (ART) cycle (in vitro fertilisation, IVF, or intracytoplasmic sperm injection, ICSI) before inclusion into the trial, where unsuccessful is defined as no embryo transfer or no pregnancy was achieved. Former ART cycles, which resulted in live birth do not count.
  3. Hypersensitivity or intolerance to pentoxifylline, xanthine derivatives or any of the excipients of the IMP.
  4. Heavy consumer of stimulating drinks (more than five cups of coffee, tea, chocolate or cola drinks per day, or more than one can [250 mL] of energy drink per day). Daily consumption of more than 24 g alcohol per day. Smoker with more than five cigarettes per day, including portions of smokeless tobacco, nicotine patches and electronic cigarettes.
  5. Any active substance abuse of drugs, medications or alcohol within the last five years.
  6. Prohibited concomitant therapies within 28 days before visit VS1 until last treatment visit:

     1. Any preparations with sex hormones or modulators of the genital system.
     2. Selective estrogen receptor modulators (SERMs), such as tamoxifen or clomifene.
     3. Aromatase inhibitors.
     4. Oral pentoxifylline.
     5. Non-medical practitioners consultations in regards to fertility.
  7. Change in intake regimen of the following therapies within 14 days before visit VS1 until last treatment visit:

     1. Herbal supplements, such as ginseng, maca or yohimbe.
     2. Dietary supplements, such as vitamins, selenium, zinc, carnitine, folic acid or coenzyme Q.
  8. Infection with human immunodeficiency virus (HIV), hepatitis B or C, genital herpes, chlamydia, gonorrhoea or syphilis.
  9. History of malignant disease (cancer). Previous or planned chemotherapy or radiotherapy.
  10. History of cerebral or retinal haemorrhage, acute myocardial infarction, severe cardiac arrhythmia or severe hepatic impairment.
  11. Family history of genetic risk factors concerning pregnancy or birth. Known abnormal karyotype.
  12. Any other condition of the subject that in the opinion of the investigator may compromise evaluation of the trial treatment or may jeopardise subject's safety, compliance or adherence to protocol requirements.
  13. Previous enrolment in this trial, or participation in any other clinical trial within the past 30 days prior to enrolment.
  14. Employees of the investigator or trial centre, with direct involvement in the proposed trial or other studies under the direction of that investigator or trial centre, as well as family members of the employees or the principal investigator.
  15. Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.

      Exclusion criteria for males:
  16. Varicocele, as confirmed by physical and ultrasound examination.

      Exclusion criteria for females:
  17. History of anovulation. History of or known current poly-cystic ovary syndrome (PCOS), endometriosis type III or IV according to the American Society for Reproductive Medicine (ASRM) criteria, or fallopian tube obstruction.
  18. Previous gynaecological surgery. One Caesarian section more than two years prior to VS1 and/or myomectomy more than 6 months prior to VS1 will be permitted.
  19. History of three or more clinical or preclinical (absence of gestational sac) miscarriages.
  20. Induced or spontaneous abortion within one year prior to VS1.
  21. Prohibited concomitant therapies within 14 days before visit VS1 until last treatment visit: Any intravaginal preparations including, but not limited to, intravaginal prescription or over-the-counter medications, vaginal lubricants, vaginal moisturizers or vaginal douches.
  22. Pregnancy or lactation.
  23. Any contraindication to becoming pregnant.
  24. Abnormal cervical smear (Bethesda classification AGC, LSIL or HSIL; PAP 3 or higher) during screening period. Cervical smear results from within the previous 12 months prior to VS1 are acceptable if the report is available to the investigator.

      Additional exclusion criterion for females at visit VR:
  25. Pregnancy.

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Efficacy assessed by rate o clinical pregnancies with fetal heart beat) of up to three treatment cycles with PKB171 vaginal gel compared to placebo vaginal gel in couples with asthenozoospermia | 9 months
  In case pregnancy was detected after the double-blind post-treatment period by a positive pregnancy test, the fetal heart activities were examined by transvaginal ultrasound (TVUS)

SECONDARY OUTCOMES:
Local IMP tolerability | 4 months
  Local IMP tolerability within 4 hours after each IMP administration up to three treatment cycles with PKB171 vaginal gel compared to placebo vaginal gel in couples with asthenozoospermia.
  Local tolerability included five parameters: Reddening, itching, burning sensation, pain, pain urination.
Safety up to three treatment cycles with PKB171 vaginal gel. | 4 months
  All AEs, including SAEs,ocurring within the period of observation for the clinical trial were recorded

CONTACTS AND LOCATIONS:
Overall Officials: José M Palacios, MD, Study Chair — Prokrea BCN, S.L.; Sara Peralta, MD, Principal Investigator — Hospital Clinic i provincial de Barcelona
Locations (1):
- José Maria Palacios, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The trial terminated prematurely due to the low number of subjects selected and high selection failure rates, despite several protocol modifications